CLINICAL TRIAL: NCT03865849
Title: Comparison of Cooled Versus Conventional Radiofrequency Treatment of the Genicular Nerves for Chronic Knee Pain: a Multicentre Randomised Controlled Non-inferiority Pilot Trial
Brief Title: Cocogen Trial: COoled Versus COnventional Radiofrequency Treatment of the GENicular Nerves for Chronic Knee Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ziekenhuis Oost-Limburg (Other)
Collaborators: Rijnstate Hospital (Other); Maastricht University Medical Center (Other)
Responsible Party: Principal Investigator, Jan Van Zundert, Principal Investigator, Ziekenhuis Oost-Limburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: COCOGEN
Record Dates: First submitted 2019-03-04; First posted 2019-03-07 (Actual); Last update posted 2023-04-13 (Actual); Status verified 2023-04

CONDITIONS: Knee Osteoarthritis
MeSH Terms: conditions — Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Prospective, multicentre, double blind, randomised controlled, non-inferiority, pilot study.
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional radiofrequent treatment (Active Comparator): The patient is placed in a supine position on a fluoroscopy table with the index knee flexed 10-15°. The procedure is performed with a 100 mm long, 18 G straight RF cannula/introducer (Halyard) with a probe/electrode with a 10 mm active tip
  Interventions: Device: Conventional radiofrequent treatment
- Cooled radiofrequent treatment (Active Comparator): The procedure is performed with a 100 mm long, 18 G straight RF cannula/introducer (Halyard) with a probe/electrode with a 100 mm long, 17 G RF cannula/introducer with an 18 G cooled probe/electrode with a 4 mm active tip (Halyard/Coolief).
  Interventions: Device: Cooled radiofrequent treatment

INTERVENTIONS:
Device: Cooled radiofrequent treatment — In the cooled radiofrequency group a treatment of 60°C measured at the tip and on average 80°C in the targeted tissue is applied during 150 seconds using the Coolief system.
  Other Names: COOLIEF™ system
  Arms: Cooled radiofrequent treatment
Device: Conventional radiofrequent treatment — In the conventional radiofrequency group a treatment of 80°C at the tip is applied during 90 seconds at each nerve.
  Arms: Conventional radiofrequent treatment

SUMMARY:
Knee osteoarthritis is a progressive degenerative process that affects joint cartilage and the subchondral bone. Approximately 10% to 30% of all osteoarthritis patients suffer from disabling symptoms such as pain, stiffness and loss of function leading to psychological and sleeping disorders and a diminished quality of life. When conservative treatment fails to treat the symptoms, a total knee arthroplasty can be performed. However, this procedure is not suitable for all patients. For these specific groups of patients a radiofrequent treatment of the genicular nerves might be an alternative treatment option. Multiple researchers investigated the effect of conventional and later also, cooled radiofrequent treatment of the genicular nerves, with promising results for both techniques. However, the techniques have never been compared in a randomised controlled trial. This study is designed to assess the feasibility of conducting a large RCT comparing pain relief and costs after a conventional radiofrequency treatment of the genicular nerves (superomedial, superolateral and inferomedial) versus a cooled radiofrequency treatment.

DETAILED DESCRIPTION:
This pilot study is designed as a prospective, multicentre, double blind, randomised controlled non-inferiority trial. The total follow up time is 6 months with follow up assessments at 1, 3 and 6 months post intervention. It is estimated that the total duration of data collection will cover 1 year. Adult patients (> 18 years) with chronic, moderate to severe knee pain (NRS>4) due to osteoarthritis, radiological diagnosed to be graded 2-4 according to the Kellgren-Lawrence criteria or with persistent postoperative moderate to severe knee pain (NRS>4) after total knee arthroplasty can be included in the study.

Patients will be randomly selected for treatment with conventional radiofrequent treatment or cooled radiofrequent treatment of the SL, SM and IL genicular nerves. In total, three hospitals participate in this study: Ziekenhuis Oost-Limburg (Belgium), Maastricht UMC+ (Netherlands) and Rijnstate (Netherlands).

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Able to understand the informed consent form and provide written informed consent and able to complete outcome measures.
* Chronic anterior knee pain (> 12 months) with an NRS > 4 on most or all days for the index knee either constantly or with motion.
* Unresponsive to conventional treatments continued during 12 months including physiotherapy, oral analgesics or intra-articular infiltrations.
* Radiologic confirmation of arthritis of OA grade of 2 (mild), 3 (moderate) or 4 (severe) noted within 6 months for the index knee according the Kellgren Lawrence criteria (27) diagnosed by an independent radiologist with experience in musculoskeletal imaging or patients with total knee arthroplasty of the index knee with a negative orthopaedic workout.
* Other therapies (including surgical interventions) for pain in the index knee are allowed for the period of the study follow up as long as they are documented. This is necessary to correctly estimate the costs in the cost effectiveness analyses. Allowing patients to receive additional treatments will also improve the protocol compliance.
* Agree to provide informed consent and to comply with the requirements of this protocol for the full duration of the study

Exclusion Criteria:

* Patient refusal to comply to protocol procedures or schedule
* Local or systemic infection (bacteraemia)
* Evidence of inflammatory arthritis or an inflammatory systemic disease responsible for knee pain
* Intra-articular injections (steroids, hyaluronic acid, platelet enriched plasma, …) in the index knee during the 3 months prior to procedure
* Body mass index (BMI) > 40 kg/m2
* Pregnant, nursing or planning to become pregnant Chronic widespread pain before the treatment
* Patients with psychosocial dysfunction will be referred for further psychological follow up prior to possible inclusion
* Allergies to products used during the procedure
* Uncontrolled coagulopathy defined as supratherapeutic dose of anticoagulation medication.
* Uncontrolled immune suppression
* Participating in another clinical trial/investigation within 30 days prior to signing informed consent
* Patient is currently implanted with a defibrillator, neuromodulator or other electrical devices
* Radicular pain in index leg
* Patient received previous conventional or cooled radiofrequency of the index knee

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2020-02-02 (Actual); Primary Completion 2021-07-28 (Actual); Study Completion 2021-10-28 (Actual)

PRIMARY OUTCOMES:
The change in pain intensity | at 1, 3, 6 and 12 months post intervention
  NRS is a unidimensional, subjective measurement of pain intensity, expressed by the patient as a number between 0 and 10. It is a 11 point scale in which 0 equals no pain and 10 maximal pain.

SECONDARY OUTCOMES:
Patient self-reported impression of change | at 1, 3, 6 and 12 months post intervention
  Patient self-reported impression of change, measured by the Patient's Global Impression of Change (PGIC). The impression of change is measured using a 7 point likert scale ranging from "very much worse (7)" to "very much improved (1)."
The change in medication use | at 1, 3, 6 and 12 months post intervention
  The change in medication use, measured by the change in Medication Quantification Scale III (MQS III). The MQS is designed as a methodology of quantifying different drug regimens in 1992 and updated in 1998 (MQS II) and 2003 (MQS III) using detriment weights determined by surveying physician members of the American Pain Society
The duration of pain relief | at 3, 6 and 12 months post intervention
  This is defined as the time interval in which a NRS reduction of more than 50% is obtained or in which the pain is still acceptable without the usage of other additional therapies (increase in MQS 3 score of more than 50%, intra-articular infiltration, operation)
The change in physical function | at baseline, 3, 6 and 12 months post intervention
  This will be measured by the change in the Oxford Knee Score (OKS). The OKS is a patient-reported measure assessing pain intensity and physical function. The list consists of 12 items scored from 1 to 5, with 0 representing normal function/ least symptoms.
The change in health-related quality of life | at baseline and at 1, 3, 6 and 12 months post intervention.
  This measured by the change in EQ-5D-5L,intervention.The EQ-5D-5L is a patient-reported generic measure of HRQoL comprising five dimensions: mobility, self-care, usual activities, pain/discomfort and anxiety/depression. Responses to the 5 items (one for each dimension) result in a patient's health state that can be transformed into a utility score ranging between 0 (death) and 1 (full health), representing the quality of life of the health state.
Hospital Anxiety and Depression Scale (HADS) | at baseline and at 1, 3, 6 and 12 months post intervention.
  HADS is developed to detect anxiety and depression in patients with physical health problems. The questionnaire consists of 14 items: 7 items to measure anxiety and 7 items to measure depression
Pain Catastrophizing Scale (PCS) | at baseline and at 1, 3 and 6 months post intervention.
  The PCS is often used in clinical settings to measure catastrophic thinking related to pain. The 13 item questionnaire consists of 3 subscales (magnification, rumination and helplessness) and asks patients to reflect on past painful experiences and to indicate the degree on which they experiences each of 13 thoughts of feelings on a 5- point scale (0 not at all and 4 all the time).
Goniometry knee | at baseline and at 3 and 6 months post intervention.
  Knee flexion and extension is assessed using a phone app meant to simulate a goniometer. The goniometry results are expressed in degrees.
Timed up and go test | at baseline and at 3 and 6 months post intervention.
  In the timed up and go test, subjects are asked to rise from a standard armchair, walk to a marker 3 m away, turn, walk back, and sit down again. The results are expressed in minutes or seconds.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Van Zundert, MD, Principal Investigator — Maastricht University Medical Centre
Locations (3):
- Ziekenhuis Oost-Limburg, Genk, Belgium
- Netherlands (2):
  - Pain Medicine Rijnstate, Arnhem
  - Pain Medicine, Maastricht University Medical Centre, Maastricht

REFERENCES:
- [Derived] Belba A, Vanneste T, Kallewaard JW, van Kuijk SM, Gelissen M, Emans P, Bellemans J, Smeets K, Van Boxem K, Sommer M, Kimman M, Van Zundert J. Cooled versus conventional radiofrequency treatment of the genicular nerves for chronic knee pain: 12-month and cost-effectiveness results from the multicenter COCOGEN trial. Reg Anesth Pain Med. 2025 Jan 7;50(1):36-45. doi: 10.1136/rapm-2023-105127. PMID 38388017
- [Derived] Vanneste T, Belba A, Kallewaard JW, van Kuijk SMJ, Gelissen M, Emans P, Bellemans J, Smeets K, Terwiel C, Van Boxem K, Sommer M, Van Zundert J. Comparison of cooled versus conventional radiofrequency treatment of the genicular nerves for chronic knee pain: a multicenter non-inferiority randomized pilot trial (COCOGEN trial). Reg Anesth Pain Med. 2023 May;48(5):197-204. doi: 10.1136/rapm-2022-104054. Epub 2023 Jan 18. PMID 36653065